CLINICAL TRIAL: NCT00887445
Title: A Double-blind, Randomized, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SLV341 in Young Healthy Male Subjects
Brief Title: First in Man Study With SLV341
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on June 25th, 2009 due to strategic decision
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S341.1.001; 2007-007196-17; 00887445
Record Dates: First submitted 2009-01-30; First posted 2009-04-24 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Diabetes
Keywords: First in Man; SLV341; diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: SLV341
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SLV341 — 5 - 1000mg once daily
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
First in man study with single and multiple rising doses with SLV341

ELIGIBILITY:
Inclusion Criteria healthy Exclusion Criteria not healthy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters: adverse event, vital signs, 12-Lead ECG, continuous lead II ECG monitoring, laboratory safety variables and physical examination. | 7 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Plasma: Cmax, tmax, AUC, t½, λz, CL/F, and Vz/F. Urine: Aeurine, fe, and CLR | 1 - 28 days
Pharmacodynamic parameters: biochemistry and 24 h Holter monitoring. | 28 days
Interaction with Midazolam | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Meuwsen, Study Director — Solvay Pharmaceuticals
Locations (1):
- S341.1.001 Site #, London, United Kingdom